CLINICAL TRIAL: NCT04621643
Title: A Multi-center Randomized Controlled Trial of Digital Cognitive Behavior Therapy for Insomnia Compared With Digital Patient Education About Insomnia in Individuals Referred to Secondary Mental Health Services in Norway
Brief Title: Digital Cognitive Behavior Therapy for Insomnia Compared With Digital Patient Education About Insomnia in Individuals Referred to Public Mental Health Services in Norway
Acronym: Norse4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Folkehelseinstituttet (Unknown); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government); University of Virginia (Other); University of California, Berkeley (Other); Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 125068
Record Dates: First submitted 2020-09-17; First posted 2020-11-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Mental Disorder; Insomnia
Keywords: Cognitive Behavioral Therapy; Patient Education; Telemedicine; Waiting Lists
MeSH Terms: conditions — Mental Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants are blinded to their group allocation, but complete blinding is not possible as the participants may understand whether they have received the active or control condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital cognitive behavioral therapy (dCBT-I) (Experimental)
  Interventions: Behavioral: digital cognitive behavioral therapy (dCBT-I)
- Patient education about sleep (PE) (Active Comparator)
  Interventions: Behavioral: Digital patient education about insomnia (PE)

INTERVENTIONS:
Behavioral: digital cognitive behavioral therapy (dCBT-I) — dCBT-I during 9 weeks. Multicomponent intervention that includes the following: psychoeducation about sleep, sleep hygiene, sleep restriction therapy, stimulus control and challenging beliefs and perception about sleep. The digital CBT-I that will be utilized in this study is named Sleep Healthy Using The internet (SHUTi). The intervention is fully automated with no contact with health care personnel, it is interactive and adapts to input from the users. It comprises of the same elements included in face-to-face CBT-I, but the user gains access to a new educational, behavioral or cognitive module each week only after completion of digital sleep diaries. dCBT-I can be accessed on computers or hand-held devices
  Arms: digital cognitive behavioral therapy (dCBT-I)
Behavioral: Digital patient education about insomnia (PE) — Control condition PE during 9 weeks. A digital patient education program that can be accessed on computers or hand-held devices. The information overlaps with that included in the dCBT-I intervention but it does not include any of the interactive features of the dCBT-I intervention and all the information is available from the moment the PE site is opened.
  Arms: Patient education about sleep (PE)

SUMMARY:
Sleep is a fundamental human need with large impact on both psychological and somatic functioning. However, for patients with mental disorders, sleep is often disturbed. Across all diagnostic groups, sleep disturbance is one of the most common and disruptive symptoms. For decades it has been assumed that the sleep disturbance these patients experience was a secondary symptom of a primary mental disorder, but recently this has changed. Experimental and clinical data now suggest that there is a reciprocal relationship between sleep disturbance and mental disorders where they perpetuate and aggravate each other. This makes sleep disturbance a potential therapeutic target in the treatment of mental disorders. Evidence emerging the last decade indicate that providing Cognitive Behavior Therapy for Insomnia (CBT-I) to patients with mental disorders not only improves sleep, but also has clinically meaningful effects on their primary mental disorder. However, a major problem has been disseminating CBT-I and few therapists are trained in this intervention. Consequently, most patients receive sleep medication although evidence clearly indicate that CBT-I is more effective and should be the treatment of choice. In this study, the investigators will use a fully automated digital version of CBT-I that might be used to treat a large number of patients while they are still on the waiting list to receive ordinary outpatient treatment in secondary mental health care clinics in Norway. The main goal is to test the effectiveness of digital CBT-I for this patient group.

DETAILED DESCRIPTION:
(27th May 2021) We have revised one of the study exclusion criteria. In the initial protocol we reported that we would exclude individuals with clinical evidence of sleep apnea, namely, we stated that: "Sleep apnea screening: An Epworth Sleepiness Scale (ESS) score >=13, indicative of high levels of objective daytime sleepiness associated with organic sleep disorders and/or positive endorsement of a screening question for sleep apnea (the item asks if they "usually or everyday snore and stop breathing and have difficulties staying awake during the day")." We have now modified the exclusion criterion, so that it is based on the screening question alone. Our updated exclusion criterion is now stated as follows: "Sleep apnea screening: A positive endorsement of a screening question for sleep apnea (the item asks if they "usually or everyday snore and stop breathing and have difficulties staying awake during the day")." i.e. the ESS score is no longer part of the assessment for eligibility for inclusion. The rationale for this change is that several publications and international experts have questioned the reliability and validity of the ESS cut-off score (>=13) when the scale is used in psychiatric outpatient populations (psychometrics in clinical samples are only modest when compared with ESS for screening community-based and/or non-clinical samples). As such ESS score is no longer used as an exclusion criterion, but we will continue to collect these data at baseline assessment and will report the ESS scores for the recruited sample.

At the time of making the amendment, 29 participants had been excluded on the basis of the ESS score.

(27th Feb, 2023): In the protocol that was approved by the Regional Committees for Medical and Health Research Ethics before inclusion started, under 'sample size', we wrote: "As the planned RCT involves limited contact between researchers and participants and has a 12-month follow-up, we have predicted that the study dropout rate is likely to reach about 50%. Therefore, we aim to recruit 800 participants, to enable us to retain 400 patients (200 in each treatment arm) at the end of the RCT."

We have now included 790 participants in this trial, and the attrition rate at the 12 month follow-up assessment is somewhat higher than predicted before we started the trial. Currently, 46% of the participants have completed the 12 month follow-up assessment. Based on this, we will not reach the target of retaining 400 participants at the end of the RCT with a sample size of 800 participants.

We have described the situation to the Regional Committees for Medical and Health Research Ethics. They have approved inclusion of new participants until June 30th 2023. This has been presented to the leaderships of the participating centers who also have approved inclusion until June 30th 2023. We will therefore recruit participants until this date. Based on our projections we will have retained at least 404 participants at the end of the RCT at this date.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Insomnia Severity Index (ISI) > 11 We have used this cut-off score previously to identify individuals who are likely to be experiencing clinical significant insomnia and who will potentially benefit from the dCBT-I intervention. Kallestad et al 2018 and a trial from Norway (Filosa et al in press) suggest that this cut-off is the most sensitive to detect a diagnosis of Insomnia Disorder.

Exclusion Criteria:

1. Sleep apnea screening: Positive endorsement of a screening question for sleep apnea (the item asks if they "usually or everyday snore and stop breathing and have difficulties staying awake during the day")
2. Medical history indicative of (i) epilepsy plus self-report of >=1 seizure <12 months ago, or (ii) recent surgery for heart disease, or (iii) currently in an attack phase of multiple sclerosis.
3. Individuals whose work schedule includes night shifts.
4. Pregnancy
5. Inadequate opportunity to sleep or circumstances prevent modification of sleep pattern (e.g. having a child aged<12 months residing home).
6. Currently receiving psychological treatment for insomnia.
7. Not a patient at one of the participating clinics.
8. Not having completed baseline assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 911 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Between-group difference in insomnia severity at week 9 after randomization | 9 weeks after randomization
  Assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.

SECONDARY OUTCOMES:
Between-group difference in insomnia severity at week 33 after randomization | 33 weeks after randomization
  While between-group difference on the ISI on week 9 is our primary endpoint, we will also assess between group differences on the ISI at week 33 (six months after post-assessment) and week 61 (one year after post assessment). Assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Between-group difference in insomnia severity at week 61 after randomization | 61 weeks after randomization
  While between-group difference on the ISI on week 9 is our primary endpoint, we will also assess between group differences on the ISI at week 33 (six months after post-assessment) and week 61 (one year after post assessment). Assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Prospective daily sleep-wake pattern at week 9 after randomization | 9 weeks after randomization
  Assessed with the Consensus Sleep Dairy, which will be completed by the participant at baseline and each follow-up point for at least 10 out of 14 consecutive days.
Prospective daily sleep-wake pattern at week 33 after randomization | 33 weeks after randomization
  Assessed with the Consensus Sleep Dairy, which will be completed by the participant at baseline and each follow-up point for at least 10 out of 14 consecutive days.
Prospective daily sleep-wake pattern at week 61 after randomization | 61 weeks after randomization
  Assessed with the Consensus Sleep Dairy, which will be completed by the participant at baseline and each follow-up point for at least 10 out of 14 consecutive days.
Chronotype at week 9 after randomization | 9 weeks after randomization
  Assessed with the Reduced Morningness - Eveningness Questionnaire (rMEQ), a widely used measure of chronotype i.e. time preference for daily activities, including bed-times. The rMEQ has five items yielding scores from 4 to 25, with lower scores indicating "eveningness" and higher scores indicating "morningness". Higher scores indicate higher levels of morningness. Scores can be divided into five categories: definitely evening type (score <8), moderately evening type (Score 8-11), neither type (score 12-17), moderately evening type (score 18-21), and definitely morning type (score >21)
Chronotype at week 33 after randomization | 33 weeks after randomization
  Assessed with the Reduced Morningness - Eveningness Questionnaire (rMEQ), a widely used measure of chronotype i.e. time preference for daily activities, including bed-times. The rMEQ has five items yielding scores from 4 to 25, with lower scores indicating "eveningness" and higher scores indicating "morningness". Higher scores indicate higher levels of morningness. Scores can be divided into five categories: definitely evening type (score <8), moderately evening type (Score 8-11), neither type (score 12-17), moderately evening type (score 18-21), and definitely morning type (score >21)
Chronotype at week 61 after randomization | 61 weeks after randomization
  Assessed with the Reduced Morningness - Eveningness Questionnaire (rMEQ), a widely used measure of chronotype i.e. time preference for daily activities, including bed-times. The rMEQ has five items yielding scores from 4 to 25, with lower scores indicating "eveningness" and higher scores indicating "morningness". Higher scores indicate higher levels of morningness. Scores can be divided into five categories: definitely evening type (score <8), moderately evening type (Score 8-11), neither type (score 12-17), moderately evening type (score 18-21), and definitely morning type (score >21)
Frequency of nightmares at week 9 after randomization | 9 weeks after randomization
  Assessed with the Nightmare Frequency Questionnaire (NFQ), a 2-item measure for frequency of nights with nightmares (in days per week, month or year) and number of nightmares (per week, month or year) an individual has experienced the last three months
Frequency of nightmares at week 33 after randomization | 33 weeks after randomization
  Assessed with the Nightmare Frequency Questionnaire (NFQ), a 2-item measure for frequency of nights with nightmares (in days per week, month or year) and number of nightmares (per week, month or year) an individual has experienced the last three months
Frequency of nightmares at week 61 after randomization | 61 weeks after randomization
  Assessed with the Nightmare Frequency Questionnaire (NFQ), a 2-item measure for frequency of nights with nightmares (in days per week, month or year) and number of nightmares (per week, month or year) an individual has experienced the last three months
Self-reported mental health status at week 9 after randomization | 9 weeks after randomization
  Assessed with the Outcome Questionnaire - 45.2 (OQ-45.2), a 45 item self-report scale for mental health status, specifically designed for patient progress throughout therapy. It has excellent internal consistency and is highly correlated with well-known outcomes such as the Symptom Checklist 90R, Beck Depression Inventory, The State Trait Inventory, The inventory of interpersonal problems, The Social Adjustment Scale, and the SF-36.34 The scale is scored on a scale of 0 (=never) to 5 (=almost always) giving a range of 0 to 180, with higher scores indicating higher levels of psychopathology. The OQ-45.2 has three validated subscales: symptom distress, interpersonal relations, and social role functioning (perceived level of difficulties in the workplace, school or home duties). Results will be reported for the sum score, and for the three subscales. The OQ-45.2 has an established clinical cut-off value and reliable change index
Self-reported mental health status at week 33 after randomization | 33 weeks after randomization
  Assessed with the Outcome Questionnaire - 45.2 (OQ-45.2), a 45 item self-report scale for mental health status, specifically designed for patient progress throughout therapy. It has excellent internal consistency and is highly correlated with well-known outcomes such as the Symptom Checklist 90R, Beck Depression Inventory, The State Trait Inventory, The inventory of interpersonal problems, The Social Adjustment Scale, and the SF-36.34 The scale is scored on a scale of 0 (=never) to 5 (=almost always) giving a range of 0 to 180, with higher scores indicating higher levels of psychopathology. The OQ-45.2 has three validated subscales: symptom distress, interpersonal relations, and social role functioning (perceived level of difficulties in the workplace, school or home duties). Results will be reported for the sum score, and for the three subscales. The OQ-45.2 has an established clinical cut-off value and reliable change index
Self-reported mental health status at week 61 after randomization | 61 weeks after randomization
  Assessed with the Outcome Questionnaire - 45.2 (OQ-45.2), a 45 item self-report scale for mental health status, specifically designed for patient progress throughout therapy. It has excellent internal consistency and is highly correlated with well-known outcomes such as the Symptom Checklist 90R, Beck Depression Inventory, The State Trait Inventory, The inventory of interpersonal problems, The Social Adjustment Scale, and the SF-36.34 The scale is scored on a scale of 0 (=never) to 5 (=almost always) giving a range of 0 to 180, with higher scores indicating higher levels of psychopathology. The OQ-45.2 has three validated subscales: symptom distress, interpersonal relations, and social role functioning (perceived level of difficulties in the workplace, school or home duties). Results will be reported for the sum score, and for the three subscales. The OQ-45.2 has an established clinical cut-off value and reliable change index
Anxiety/depression at week 9 after randomization | 9 weeks after randomization
  Assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire for non-vegetative symptoms of anxiety and depression on a 0 to 3 likert scale. The sum score can be used as a measure of general psychological distress and is widely used in the community, general practice and psychiatric settings. It has a range of 0 to 42 points with higher scores indicating higher levels of psychological distress.
Anxiety/depression at week 33 after randomization | 33 weeks after randomization
  Assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire for non-vegetative symptoms of anxiety and depression on a 0 to 3 likert scale. The sum score can be used as a measure of general psychological distress and is widely used in the community, general practice and psychiatric settings. It has a range of 0 to 42 points with higher scores indicating higher levels of psychological distress.
Anxiety/depression at week 61 after randomization | 61 weeks after randomization
  Assessed with the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire for non-vegetative symptoms of anxiety and depression on a 0 to 3 likert scale. The sum score can be used as a measure of general psychological distress and is widely used in the community, general practice and psychiatric settings. It has a range of 0 to 42 points with higher scores indicating higher levels of psychological distress.
Fatigue at week 9 after randomization | 9 week after randomization
  Assessed with the Chalder Fatigue Scale (CFS), a 11-item questionnaire for daytime physical and psychological fatigue on a 0 to 3 likert scale (0=less than usual, 3=much more than usual). The scale has a range of 0 to 33 with higher scores indicating higher levels of fatigue. Two additional items assess duration of fatigue (0=less than a week, 4=six months or more) and how much of the time the individual experience fatigue (0=25% of the time, 3=all the time)
Fatigue at week 33 after randomization | 33 weeks after randomization
  Assessed with the Chalder Fatigue Scale (CFS), a 11-item questionnaire for daytime physical and psychological fatigue on a 0 to 3 likert scale (0=less than usual, 3=much more than usual). The scale has a range of 0 to 33 with higher scores indicating higher levels of fatigue. Two additional items assess duration of fatigue (0=less than a week, 4=six months or more) and how much of the time the individual experience fatigue (0=25% of the time, 3=all the time)
Fatigue at week 61 after randomization | 61 weeks after randomization
  Assessed with the Chalder Fatigue Scale (CFS), a 11-item questionnaire for daytime physical and psychological fatigue on a 0 to 3 likert scale (0=less than usual, 3=much more than usual). The scale has a range of 0 to 33 with higher scores indicating higher levels of fatigue. Two additional items assess duration of fatigue (0=less than a week, 4=six months or more) and how much of the time the individual experience fatigue (0=25% of the time, 3=all the time)
General health state at week 9 after randomization | 9 weeks after randomization
  Assessed with Euroqol-5D, a 5-item self-report questionnaire for general health state on a 0 to 5 likert scale. It measures levels of problems with walking, performing self-care, doing usual activities, pain/discomfort, and anxiety/depression. It is widely used across Europe in assessments of health resources utilization as it allows measurement of Quality Adjusted Life Years (QALYs) in individuals presenting with a wide range of physical and mental disorders
General health state at week 33 after randomization | 33 weeks after randomization
  Assessed with Euroqol-5D, a 5-item self-report questionnaire for general health state on a 0 to 5 likert scale. It measures levels of problems with walking, performing self-care, doing usual activities, pain/discomfort, and anxiety/depression. It is widely used across Europe in assessments of health resources utilization as it allows measurement of Quality Adjusted Life Years (QALYs) in individuals presenting with a wide range of physical and mental disorders
General health state at week 61 after randomization | 61 weeks after randomization
  Assessed with Euroqol-5D, a 5-item self-report questionnaire for general health state on a 0 to 5 likert scale. It measures levels of problems with walking, performing self-care, doing usual activities, pain/discomfort, and anxiety/depression. It is widely used across Europe in assessments of health resources utilization as it allows measurement of Quality Adjusted Life Years (QALYs) in individuals presenting with a wide range of physical and mental disorders
Frequency of alcohol use at week 9 after randomization | 9 weeks after randomization
  Assessed with the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a three-item self-report questionnaire assessing frequency of alcohol use (0=never, 4=four times each week or more), number of units typical for a drinking day (0=1-2 units, 4=10 or more units), and frequency of binge-drinking (0=never, 4=daily or almost daily). It is a short-version of the 10-item AUDIT developed by the World Health Organization
Frequency of alcohol use at week 33 after randomization | 33 weeks after randomization
  Assessed with the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a three-item self-report questionnaire assessing frequency of alcohol use (0=never, 4=four times each week or more), number of units typical for a drinking day (0=1-2 units, 4=10 or more units), and frequency of binge-drinking (0=never, 4=daily or almost daily). It is a short-version of the 10-item AUDIT developed by the World Health Organization
Frequency of alcohol use at week 61 after randomization | 61 weeks after randomization
  Assessed with the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a three-item self-report questionnaire assessing frequency of alcohol use (0=never, 4=four times each week or more), number of units typical for a drinking day (0=1-2 units, 4=10 or more units), and frequency of binge-drinking (0=never, 4=daily or almost daily). It is a short-version of the 10-item AUDIT developed by the World Health Organization
Headache impact at week 9 after randomization | 9 weeks after randomization
  Assessed with the Headache Impact Test - 6 (HIT-6), a six-item self-report questionnaire assessing intensity and consequences of headaches the last month, rated from never to always. The scale has a range from 36 to 78 with higher values indicating higher severity of headaches.
Headache impact at week 33 after randomization | 33 weeks after randomization
  Assessed with the Headache Impact Test - 6 (HIT-6), a six-item self-report questionnaire assessing intensity and consequences of headaches the last month, rated from never to always. The scale has a range from 36 to 78 with higher values indicating higher severity of headaches.
Headache impact at week 61 after randomization | 61 weeks after randomization
  Assessed with the Headache Impact Test - 6 (HIT-6), a six-item self-report questionnaire assessing intensity and consequences of headaches the last month, rated from never to always. The scale has a range from 36 to 78 with higher values indicating higher severity of headaches.
Work performance in daily living at week 9 after randomization | 9 weeks after randomization
  Assessed with the Work Productivity and Impairment Questionnaire General Health (WPAI:GH) for work performance and impairment in daily living. It is a six-item questionnaire that measures: sickness absenteeism; sickness presenteeism; overall work impairment and; activity impairment.
Work performance in daily living at week 33 after randomization | 33 weeks after randomization
  Assessed with the Work Productivity and Impairment Questionnaire General Health (WPAI:GH) for work performance and impairment in daily living. It is a six-item questionnaire that measures: sickness absenteeism; sickness presenteeism; overall work impairment and; activity impairment.
Work performance in daily living at week 61 after randomization | 61 weeks after randomization
  Assessed with the Work Productivity and Impairment Questionnaire General Health (WPAI:GH) for work performance and impairment in daily living. It is a six-item questionnaire that measures: sickness absenteeism; sickness presenteeism; overall work impairment and; activity impairment.
Subjective cognitive disfunction at week 9 after randomization | 9 weeks after randomization
  Assessed with the Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA), a 16-item self-reported instrument of subjective cognitive dysfunctions including executive function, processing speed, working memory, verbal learning and memory, attention/concentration and mental tracking. Items are rated using a 4-point scale. The higher the score, the more subjective complaints. Although the assessment was initially introduced for use with individuals with bipolar disorders, the rating can be used ion other clinical populations
Subjective cognitive disfunction at week 33 after randomization | 33 weeks after randomization
  Assessed with the Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA), a 16-item self-reported instrument of subjective cognitive dysfunctions including executive function, processing speed, working memory, verbal learning and memory, attention/concentration and mental tracking. Items are rated using a 4-point scale. The higher the score, the more subjective complaints. Although the assessment was initially introduced for use with individuals with bipolar disorders, the rating can be used ion other clinical populations
Subjective cognitive disfunction at week 61 after randomization | 61 weeks after randomization
  Assessed with the Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA), a 16-item self-reported instrument of subjective cognitive dysfunctions including executive function, processing speed, working memory, verbal learning and memory, attention/concentration and mental tracking. Items are rated using a 4-point scale. The higher the score, the more subjective complaints. Although the assessment was initially introduced for use with individuals with bipolar disorders, the rating can be used ion other clinical populations
Opinion on negative effects of the intervention at week 9 after randomization | 9 weeks after randomization
  Assessed with the Negative Effects Questionnaire (NEQ), a self-report measure that contains 20 items that are scored on a five-point Likert-scale (rated 0-4) where higher scores indicate higher levels of negative effects. After each item, the individual is asked whether they consider the effect to be caused by the intervention received or caused by other circumstances (yes/no), as well as one open-ended question
Impact on future treatment at week 9 after randomization | 9 weeks after randomization
  This will be assessed post intervention with two items. The first will assess if this intervention has impacted motivation for face-to-face treatment for mental disorders, the second will assess if this intervention has impacted motivation for specifically working with sleep interventions at a later time (both scored on a 1 to 9 scale with 1=very unmotivated, 9=very motivated)
Use of therapeutic techniques at week 9 after randomization | 9 weeks after randomization
  Assessed with the Use of Sleep Strategies (USS), a six item self-report questionnaire developed to measure how often individuals use six different therapeutic techniques (keep a stable rise time, refrain from sleeping during daytime, use the bed and bedroom only for sleeping, practiced sleep restriction, practiced stimulus control) and their perception of its utility. The techniques are integral to CBT-I but are also described in sleep psychoeducation or hygiene programmes
Use of therapeutic techniques at week 33 after randomization | 33 weeks after randomization
  Assessed with the Use of Sleep Strategies (USS), a six item self-report questionnaire developed to measure how often individuals use six different therapeutic techniques (keep a stable rise time, refrain from sleeping during daytime, use the bed and bedroom only for sleeping, practiced sleep restriction, practiced stimulus control) and their perception of its utility. The techniques are integral to CBT-I but are also described in sleep psychoeducation or hygiene programmes
Use of therapeutic techniques at week 61 after randomization | 61 weeks after randomization
  Assessed with the Use of Sleep Strategies (USS), a six item self-report questionnaire developed to measure how often individuals use six different therapeutic techniques (keep a stable rise time, refrain from sleeping during daytime, use the bed and bedroom only for sleeping, practiced sleep restriction, practiced stimulus control) and their perception of its utility. The techniques are integral to CBT-I but are also described in sleep psychoeducation or hygiene programmes
Insomnia symptoms and severity at week 9 after randomization | 9 weeks after randomization
  Assessed with the Bergen Insomnia Scale (BIS). BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IVTR (American Psychiatric Association).
Insomnia symptoms and severity at week 33 after randomization | 33 weeks after randomization
  Assessed with the Bergen Insomnia Scale (BIS). BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IVTR (American Psychiatric Association).
Insomnia symptoms and severity at week 61 after randomization | 61 weeks after randomization
  Assessed with the Bergen Insomnia Scale (BIS). BIS comprises six items that assesses symptoms of insomnia based on the insomnia criteria found in the Diagnostic and Statistical Manual of Mental Disorders-IVTR (American Psychiatric Association).
Use of health care services over the 12 month trial period | From 2 years before randomization to one year follow-up
  Number of appointments at mental health care clinics, type and timing of treatment and admissions, and date of the first appointment for each patient during the study period from the Norwegian Patient Registry. Longer term follow-up (>12 month) may be undertaken.
Medication use at baseline over the 12 month trial period | From 2 years before randomization to one year follow-up
  Dose, timing, and type of prescribed hypnotic, sedative/anxiolytic, antidepressant and other psychotropic medications (According to the WHO Anatomical Therapeutic Chemical Classification System) and changes recorded during the RCT (data from the Norwegian Prescription Database). Longer term follow-up (>12 month) may be undertaken.
Costs of treatment offered by the public services over the 12 month trial period | From 2 years before randomization to one year follow-up
  Data from the database named 'Kontroll og Utbetaling av Helserefusjon'. Longer term follow-up (>12 month) may be undertaken.
Sick leave or in receipt of disability benefits over the 12 month trial period | From 2 years before randomization to one year follow-up
  Data from the administrative database called Forløpsdatabasen. Longer term follow-up (>12 month) may be undertaken.
Cause of death | From baseline to 12 month follow-up
  Data about the cause of death from the database called "Dødsårsaksregisteret". Longer term follow-up (>12 month) may be undertaken

CONTACTS AND LOCATIONS:
Overall Officials: Pål Sandvik, md, Study Director — St Olavs Hospital, Division of Mental Health Care; Håvard Kallestad, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (4):
- Norway (4):
  - Helse Møre og Romsdal HF, Ålesund
  - AHUS, Oslo
  - Stavanger Universitetssykehus, Stavanger
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data that underlie the results will be available after publication of the final version of the trial to researchers from accredited research institutions. Access to data will be limited to investigators who provide a methodologically sound proposal and will be for a specified time period (commencing about 3 months after publication and ending after five years). To ensure GDPR compliance, data processing must be covered by the 'Standard Contractual Clauses' from the European Commission, that data requesters have to sign. Proposals and requests for data access should be directed to the principal investigator.

REFERENCES:
- [Derived] Kallestad H, Saksvik S, Vedaa O, Langsrud K, Morken G, Lydersen S, Simpson MR, Dorheim SK, Holmoy B, Selvik SG, Hagen K, Stiles TC, Harvey A, Ritterband L, Sivertsen B, Scott J. Digital cognitive-behavioural therapy for insomnia compared with digital patient education about insomnia in individuals referred to secondary mental health services in Norway: protocol for a multicentre randomised controlled trial. BMJ Open. 2021 Jun 28;11(6):e050661. doi: 10.1136/bmjopen-2021-050661. PMID 34183350